CLINICAL TRIAL: NCT02021331
Title: The Effect of Immediate Implant Placement and Provisionalization in The Esthetic Zone: A Randomized Clinical Trial
Brief Title: The Effect of Immediate Implant Placement and Provisionalization in the Esthetic Zone
Acronym: 3i
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment so sponsor stopped funding the study (did not renew)
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Robert M. Eber, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00041254
Record Dates: First submitted 2013-12-13; First posted 2013-12-27 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Jaw, Edentulous, Partially
Keywords: jaw, edentulous, partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- immediate implant placement without provisionalization (Active Comparator): The subject will have the tooth removed and an implant placed right away. In this arm the subject will have no temporary crown on the implant.
  Interventions: Device: immediate implant placement without provisionalization
- immediate implant placement with immediate provisionalization (Experimental): The subject will have the tooth removed and an implant placed right away. In this arm the subject will get a temporary crown on the implant.
  Interventions: Device: immediate implant placement with immediate provisionalization

INTERVENTIONS:
Device: immediate implant placement without provisionalization
  Other Names: BIOMET 3i Prevail Nanotite Certain - dental implant; Encode abutment
  Arms: immediate implant placement without provisionalization
Device: immediate implant placement with immediate provisionalization
  Other Names: BIOMET 3i Prevail Nanotite Certain - dental implant; Encode abutment
  Arms: immediate implant placement with immediate provisionalization

SUMMARY:
The purpose of this study is to compare two different techniques of placing dental implants: 1) removing the tooth and placing the implant immediately and 2) removing the tooth and placing both the implant and a temporary crown immediately. Both procedures currently are accepted methods for replacing missing teeth but direct comparisons of the two procedures are lacking. The results of this study should aid clinicians in selecting the best implant placement technique for their patients.

DETAILED DESCRIPTION:
To qualify, patients must be between 18 to 79 years old, in good health, have a tooth in the upper jaw (except molars) that needs to be extracted, and able and willing to return to the University of Michigan Dental School for all follow-up appointments (8 follow-up visits over a period of 12 months). Sufficient number of natural teeth and/or replacements to provide a stable occlusion as determined by the investigator

Patients will be excluded for any of the following conditions: Women who are pregnant or plan to become pregnant, an existing implant adjacent to the area of study, current smoker or quit smoking less than one year ago, antibiotic therapy for more than two weeks within 3 months of baseline, need for antibiotics prior to dental treatment (due to prosthetic joint replacement or other medical condition), chronic use of medications known to affect the gum tissues (calcium channel blocker (less than 6 months, or over 6 months and have experienced overgrowth of your gums), anticonvulsants, immunosuppressive drugs, nonsteroidal anti-inflammatory medications...), current orthodontic treatment, or active periodontal treatment. Participants must inform the investigators if they are enrolled in any other studies because it may becloud them from participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* between 18 to 79 years old
* in good health
* have a single tooth in the upper jaw (except molars) that needs to be extracted
* able and willing to return to the University of Michigan Dental School for all follow-up appointments (8 follow-up visits over a period of 12 months)
* Sufficient number of natural teeth and/or replacements to provide a stable occlusion as determined by the investigator

Exclusion Criteria:

* an existing implant adjacent to the area of study
* current smoker or quit smoking less than one year ago
* antibiotic therapy for more than two weeks within 3 months of baseline, need for antibiotics prior to dental treatment (due to prosthetic joint replacement or other medical condition)
* chronic use of medications known to affect the gum tissues (calcium channel blocker (less than 6 months, or over 6 months and have experienced overgrowth of your gums), anticonvulsants, immunosuppressive drugs, nonsteroidal anti-inflammatory medications...)
* current orthodontic treatment, or active periodontal treatment
* Women who are pregnant or plan to become pregnant during the course of the study, and nursing mothers
* unstable medical condition or if you are unable to have routine dental surgery then you should not participate in this study. If you are already participating in another study, we ask that you inform the investigators because participating in more than one study may be harmful to you.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Implant Placement Without Provisionalization: The subject will have the tooth removed and an implant placed right away. In this arm the subject will have no temporary crown on the implant.
  immediate implant placement without provisionalization
- Immediate Implant Placement With Immediate Provisionalization: The subject will have the tooth removed and an implant placed right away. In this arm the subject will get a temporary crown on the implant.
  immediate implant placement with immediate provisionalization
Period: Overall Study
Arm/Group | Immediate Implant Placement Without Provisionalization | Immediate Implant Placement With Immediate Provisionalization
Started | 2 | 3
Completed | 2 | 1
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Implant Placement Without Provisionalization | Immediate Implant Placement With Immediate Provisionalization | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Soft Tissue Diemensional Change
Description: Tissue thickness will be measured from the digital impression and CBCT data from the hard tissue.
Time Frame: Baseline, 12mo after baseline
Population: Data was not collected.
Arm/Group | Immediate Implant Placement Without Provisionalization | Immediate Implant Placement With Immediate Provisionalization
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Implant Survival
Description: Checking to make sure the implant is stable.
Time Frame: 2wk, 4wk, 6wk, 3mo, 6mo, 12mo
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Implant Placement Without Provisionalization | Immediate Implant Placement With Immediate Provisionalization
Number analyzed (Participants) | 2 | 3
Participants
  2wk | 2 | 3
  4wk | 2 | 2
  6wk | 2 | 1
  3mo | 2 | 1
  6mo | 2 | 1
  12mo | 2 | 1

3. Other Pre Specified Outcome: Bony Dimensional Changes
Description: Measurements will be based off of standardized x-rays and CBCT.
Time Frame: Baseline, 6mo & 12mo after baseline
Population: Data was not collected
Arm/Group | Immediate Implant Placement Without Provisionalization | Immediate Implant Placement With Immediate Provisionalization
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Immediate Implant Placement Without Provisionalization | Immediate Implant Placement With Immediate Provisionalization
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Implant Placement Without Provisionalization (N=2) | Immediate Implant Placement With Immediate Provisionalization (N=3)
Implant failure (Surgical and medical procedures) | 0 (0) | 2 (2)
Implant crown came off (General disorders) | 1 (1) | 0 (0)
UTI (General disorders) | 0 (0) | 1 (1)
Sinus Pain (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No